CLINICAL TRIAL: NCT04906187
Title: Impact of Specific Monitoring of Intraoperative Analgesia Under General Anesthesia on Chronic Pain After Ovarian Cancer Surgery. The MONIALC Study.
Brief Title: Impact of Specific Monitoring of Intraoperative Analgesia Under General Anesthesia on Chronic Pain After Ovarian Cancer Surgery
Acronym: MONIALC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IB 2020-04; 2020-A02767-32 (Other: ANSM IDRCB number)
Record Dates: First submitted 2021-05-20; First posted 2021-05-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Neoplasm
Keywords: ovarian neoplasm; analgesia monitoring; pain measurement; Analgesia Nociception Index
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : Experimental group with intraoperative ANI monitoring of nociception (Experimental)
  Interventions: Other: Arm A : intraoperative ANI monitoring of nociception
- Arm B : Control group without ANI intraoperative monitoring of nociception (Other)
  Interventions: Other: Arm B : no specific monitoring of nociception

INTERVENTIONS:
Other: Arm A : intraoperative ANI monitoring of nociception — For the experimental group (arm A), the sufentanil doses are adjusted to maintain an ANI between 50 and 70. Morphine doses are adjusted from 0.05 to 0.05 µg / ml. Intraoperative data will be collected for ANI, TIVA and hemodynamics.
  Arms: Arm A : Experimental group with intraoperative ANI monitoring of nociception
Other: Arm B : no specific monitoring of nociception — For the control group (arm B), adjustments to the opioid doses are made in relation to the hemodynamic reactions of the patient and the operating times. Intraoperative data will be collected for TIVA and hemodynamics.
  Arms: Arm B : Control group without ANI intraoperative monitoring of nociception

SUMMARY:
This is a single-center, randomized, phase II, non-comparative, single-blind clinical study that will determine whether morphine reduction through intraoperative monitoring by ANI (Analgesia Nociception Index) significantly reduces chronic post-surgical pain at three months after laparotomy for ovarian carcinoma with regard to standard care.

DETAILED DESCRIPTION:
Prior to carrying out the research, the informed consent of the person must be obtained after being informed of the purpose of the research, its conduct and duration, benefits, potential risks and constraints of the study.

Before inclusion,all eligibility criteria will be verified, VAS pain score and VAS anxiety will be performed.

The surgical procedure for ovarian carcinoma will be performed by laparotomy and the intraoperative monitoring of nociception wil depend of the randomization arm : Intraoperative ANI monitoring of nociception (experimental arm) versus no specific monitoring of nociception (control arm). The total dose of opioids (in micrograms) received by the patients will be recorded at the end of the surgery.

VAS pain score will be performed immediately postoperatively and at three months after the intervention. A DN4 questionnaire (neuropathic pain) will be evaluated at three months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged 18 years and over.
2. Histologically proven or strongly suspected ovarian carcinoma.
3. Indication for laparotomy surgery with xyphopubic incision.
4. Acceptance of epidural anesthesia.
5. Pain score ≤ 3 (VAS or Numeric Verbal Scale).
6. Free and informed consent.
7. Patient affiliated with a French social security scheme in accordance with French law on research involving human participants.

Exclusion Criteria:

1. Heart rhythm disturbances.
2. History of Cerebral Vascular Accident (CVA).
3. History of epilepsy.
4. Wearing a pacemaker.
5. Receiving morphine treatment preoperatively.
6. Medical contraindication to an epidural.
7. Patient unable to follow and adhere to trial procedures for geographic, social or psychological reasons.
8. Patient placed under guardianship or curatorship.
9. Patient already included in the present study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a pain score on the self-assessment VAS > 4, three months after the surgery. | 3 months after surgery
  The Visual Analog Scale (VAS) is a validated, reliable and reproducible tool. The VAS will be used to measure pain. This self-assessment scale allows the patient to evaluate his or her pain from 0 to 10 "0=No pain" to "10=Maximum imaginable pain ". A pain VAS score of 4 and above is considered clinically significant.

SECONDARY OUTCOMES:
Arm A : total dose of opioids received intraoperatively | Surgery
Arm B : total dose of opioids received intraoperatively | Surgery
Arm A : Patients' pain score on the VAS immediately postoperatively | within one hour of extubation
  The Visual Analog Scale (VAS) is a validated, reliable and reproducible tool. The VAS will be used to measure pain. This self-assessment scale allows the patient to evaluate his or her pain from 0 to 10 "0=No pain" to "10=Maximum imaginable pain ". A pain VAS score of 4 and above is considered clinically significant.
Arm B : Patients' pain score on the VAS immediately postoperatively | within one hour of extubation
  The Visual Analog Scale (VAS) is a validated, reliable and reproducible tool. The VAS will be used to measure pain. This self-assessment scale allows the patient to evaluate his or her pain from 0 to 10 "0=No pain" to "10=Maximum imaginable pain ". A pain VAS score of 4 and above is considered clinically significant.
Arm A : proportion of patients with a DN4 questionnaire score> 4, three months after surgery | 3 months after surgery
Arm B : Arm A : proportion of patients with a DN4 questionnaire score> 4, three months after surgery | 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No